CLINICAL TRIAL: NCT01912001
Title: Virtual Ward for Home Dialysis - A Novel Model to Address Transitions of Care
Brief Title: Virtual Ward for Home Dialysis
Acronym: Virtual Ward
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christopher Chan (Other)
Collaborators: Baxter Healthcare Corporation (Industry); Vancouver General Hospital (Other); Sunnybrook Health Sciences Centre (Other); St. Paul's Hospital, Canada (Other); University of Alberta (Other); Unity Health Toronto (Other); The Ottawa Hospital (Other); Capital Health Nova Scotia (Unknown)
Responsible Party: Sponsor-Investigator, Christopher Chan, Deputy Director-Nephrology/UHN, University Health Network, Toronto
Organization: University Health Network, Toronto (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 12-5397-AE
Record Dates: First submitted 2013-07-22; First posted 2013-07-30 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: End Stage Renal Disease; Kidney Failure; Home Dialysis
Keywords: end stage renal disease; kidney failure; home dialysis; hemodialysis; peritoneal dialysis; gaps in care; co-morbidity; transitions of care settings
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Telephone follow-up. (Other): A member of the Home Dialysis team will telephone patients to follow-up on their symptoms, dialysis and care.
  Interventions: Other: Telephone follow-up; Other: Sympton Assessment

INTERVENTIONS:
Other: Telephone follow-up
Other: Sympton Assessment

SUMMARY:
Home based renal replacement therapy (RRT), including peritoneal dialysis (PD) and home hemodialysis(HHD), offers enhanced quality of life and clinical advantages compared to conventional in-center hemodialysis. Patients with end stage renal disease, that is failure of the kidneys such that dialysis is required, are at high risk for adverse health events especially during a period of transition following a change in care settings. The investigators aim to implement a Home Dialysis Virtual Ward (HDVW) strategy of telephone follow-up, which is targeted to minimize gaps of care during transitions in care.

The investigators aim to have clinicians follow patients by telephone if they meet one of the following four criteria;

1. Discharge from hospital.
2. Having an interventional procedure.
3. Prescription of an antibiotic.
4. Completion of Home Dialysis training.

The major goal of this HDVW initiative is to provide appropriate and effective supports to medically complex patients in a targeted window of vulnerability.

DETAILED DESCRIPTION:
End stage renal disease (ESRD) is kidney disease that requires dialysis or kidney transplant to replace lost kidney function. The most common renal replacement therapy in North America is conventional, in-center hemodialysis (CHD). Home dialysis - including peritoneal dialysis (PD) and home hemodialysis(HHD)offers benefits to quality of life, patient satisfaction and clinical advantages, including better survival compared to CHD. (references 1-11 in the protocol).

Patients with (ESRD) have a high burden of co-morbidity. Periods of transition of care from acute care to other settings are thought to represent times of increased vulnerability. Since patients who require home dialysis have high co-morbidity and have complex medical care issues, the investigators seek to improve transitions of care for these patients with a novel strategy of follow-up.

When patients have been hospitalized, had treatment for an infection, had a procedure, or have just transitioned to home dialysis therapy,the investigators aim to decrease gaps in care by having a clinician follow-up by telephone with these patients in a scheduled way.

During the telephone call the clinician will assess the patients care and symptoms, and make adjustments to prescriptions of medications and dialysis, or referrals to additional care as required. Evaluation of care will include:

1. Indication for admission to the Virtual Ward.
2. Dialysis prescription.
3. Demographic and comorbidity data.
4. Medication reconciliation.
5. Symptom Assessment.
6. Dietary review.

Symptoms will be evaluated using a standardized patient assessment tool,the Charlson Comorbidity Index and the modified Edmonton Symptom Assessment Scale.

At the end of the Virtual Ward follow-up period, patients will be asked to complete a Patient Satisfaction Questionnaire.

Data from a preliminary vanguard pilot phase of 84 assessments done in 21 patients over 2 months indicates that 170 to 200 patients recruited from eight sites during a 10 month period should be sufficient to allow analysis of the data collected.

Each of the participating Investigator's will have input into the study conduct and publication preparation.

ELIGIBILITY:
Inclusion Criteria:

* Patient in the home dialysis program (PD and HHD)and on of the following:
* Discharge from hospital following an inpatient admissions
* Medical procedure (e.g. vascular access procedure).
* Treatment with antibiotics.
* Completion of home dialysis training program.

Exclusion Criteria:

* Decline consent.
* Unable to participate - (e.g. no phone at home, language barrier)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2013-09; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
The number of care gaps identified. | Up to 24 weeks post discharge from the virtual ward.

SECONDARY OUTCOMES:
Dialysis prescription and adherence. | Up to 24 weeks.
  Orders for dialysis treatment and amount of dialysis performed will be recorded.
Morbidity associated with dialysis therapy. | Up to 24 weeks post discharge from the virtual ward.
  All deaths will be recorded.
Burden associated with travel time for patients. | Up to 24 weeks post discharge from the virtual ward.
  Travel time for health related visits will be recorded.
Medication reconciliation. | Up to 24 weeks post discharge from the virtual ward.
  Best possible medication history will be recorded at each interaction.
Symptom management. | Up to 24 weeks post discharge from the virtual ward.
  Symptom assessment will be done at each interaction.
Adherence with dietary recommendations. | Up to 24 weeks post discharge from the virtual ward.
  Diet review will be performed at each visit.
Coordination of care among participating providers. | During virtual ward follow-up.
  Referrals and consultations will be tracked.
Patient satisfaction. | 24 weeks post discharge from the virtual ward.
  A satisfaction questionnaire will be mailed to participants at the end of participation.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher T Chan, MD, Principal Investigator — University Health Network, Toronto
Locations (7):
- Canada (7):
  - University of Alberta, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Capital District Health Authority, Halifax, Nova Scotia
  - The Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - University Health Network, Toronto, Ontario

REFERENCES:
- [Derived] Schachter ME, Bargman JM, Copland M, Hladunewich M, Tennankore KK, Levin A, Oliver M, Pauly RP, Perl J, Zimmerman D, Chan CT. Rationale for a home dialysis virtual ward: design and implementation. BMC Nephrol. 2014 Feb 14;15:33. doi: 10.1186/1471-2369-15-33. PMID 24528505